CLINICAL TRIAL: NCT04605328
Title: Cesarean Scar Defect (CSD); Prevalence, Risk Factors And Possible Associated Symptoms: A Cohort Observational Study
Brief Title: Cesarean Scar Defect (CSD); Prevalence, Risk Factors And Possible Associated Symptoms
Acronym: isthmocele
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Bahaa, Principle Investigator, Assiut University
Other Study IDs: Cesarean scar defect
Record Dates: First submitted 2020-10-05; First posted 2020-10-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Cesarean Section Complications
Keywords: niche

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Two dimension and three dimension ultrasound — Patient will undergo 2D and 3D ultrasound evaluation after CS for detection of CSD

SUMMARY:
The study aims to detect the incidence of Cesarean Scar Defect (CSD) in women undergoing CS in Women Health Hospital (WHH), assiut University, to identify risk factors for development of CSD and identify the possible gynaecological symptoms related to CSD.

DETAILED DESCRIPTION:
All eligible women, who will undergo CS in Women Health Hospital (WHH) will be seen on regular visits to detect the presence of CSD by ultrasound and identify its characters and a questionnaire will be fulfilled by the candidates about the gynecological symptoms related to CSD and appeared after CS.

ELIGIBILITY:
Inclusion Criteria:

* All women who will undergo transverse lower segment cesarean section after 28 weeks gestational age (electively and Emergency), after counseling and written consent

Exclusion Criteria:

1. Rupture uterus (unscarred or scarred).
2. Upper segment CS.
3. Vertical lower segment CS.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Women Health Hospital for performing CS will be seen on regular visits for ultrasound scan for detection of CSD
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of CSD in Women health Hospital | 1 year
  the incidence of CSD in Women health Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ayman shamaash, PHD, Study Director — Assiut University; Sherif Badran, MD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided